CLINICAL TRIAL: NCT02030236
Title: CAERvest® - A Novel Endothermic Hypothermic Device for Core Body Cooling. Safety and Efficacy Testing.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bodychillz Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAERvest-001
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Hypothermia.
Keywords: hypothermia, induced; rewarming; therapeutic; heart arrest; asystole; frostbite
MeSH Terms: conditions — Hypothermia; Heart Arrest; Frostbite | interventions — Cool-Down Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cooling (Experimental)
  Interventions: Device: Cooling

INTERVENTIONS:
Device: Cooling — Temperature reached Duration of exposure to cold.
  Other Names: CAERvest prototype

SUMMARY:
Cooling the whole body to 32-34 degrees Centigrade from the normal of around 37 degrees Centigrade for 24 hours has been shown to be an effective way of reducing damage to brain function after return of spontaneous circulation when someone has been resuscitated from cardiac arrest. Cardiac arrest is a form of heart attack where the heart stops pumping.

The device is a prototype cooling vest. The investigators anticipate that this will be useful in ambulances, helicopters and emergency departments where there is a need for a portable, safe, easy-to-use, inexpensive, external, effective, readily-controlled and single-patient use device able to reduce body temperature by at least 1 degree Centigrade an hour to initiate cooling. What the investigators are doing in these trials is to demonstrate that the investigators can cool people and to get the best design possible for patient use. That means some of the initial prototypes will not resemble what we expect the eventual device to look like. The investigators will be undertaking the initial trials on 30 normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

Human volunteers aged over 18. The upper age limit, as is standard for risk mitigation in such studies, is 35. The volunteer must have capacity to understand the trial and give informed consent to participate. If the volunteer's first language is not English we will make use of Sussex Interpreting Services, a professional interpreting service.

Exclusion Criteria:

Pregnancy. Any disclosed medical condition. Any medical condition detected on examination. Core temperature outside stated parameters.

We will ask the volunteer to confirm that they are otherwise healthy, taking no regular medication (except the oral contraceptive pill), are not using recreational drugs and have no significant past medical history, in particular cardiovascular disease of any sort, thyroid disease, diabetes mellitus or other metabolic disease.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in core body temperature by 1 degree Centigrade. | 1 hour.
  The cooling properties of the vest are under investigation, and this reduction is the primary outcome measure.

SECONDARY OUTCOMES:
Skin condition. | 3 days.
  As the cooling is performed by a cold vest applied directly to the skin we need to ensure that no skin damage is caused.
ECG abnormalities. | 3 hours.
  ECG abnormalities: ECG abnormalities are common after cardiac arrest, and have been noted in cooled patients after cardiac arrest. We will monitor the ECG for any abnormalities. The following will be noted but will not terminate the study:
  Bradycardia of less than 15 beats per minute below baseline. Unifocal ventricular ectopics. Unifocal atrial ectopics. Any other cardiac abnormality will cause immediate termination of the study and intervention to treat as necessary. A defibrillator will be available in the study room.
Sepsis. | 3 days.
  Sepsis: Increased rates of sepsis have been seen in intensive care units in patients who have received therapeutic hypothermia. We will enquire about sepsis symptoms in our follow-up contact.
Skin condition. | 3 days.
  Our aim is not to cause any skin damage to patients or volunteers. We will therefore inspect the skin after removing the vest or at any time before that if the volunteer expresses concern. We expect pallor of the skin during cooling and reddening during rewarming with some numbness and some discomfort, both during cooling and rewarming. We will regard any evidence of frostbite as a serious untoward injury (SUI) and this will result in suspension of the study and an investigation into the specific vest used and the general vest design and formulation. We regard this as a serious risk but highly unlikely in practice.

CONTACTS AND LOCATIONS:
Overall Officials: Rowland L Cottingham, FRCS FCEM, Principal Investigator — Brighton and Sussex Universities Hospital NHS Trust
Locations (1):
- CIRU, Royal Sussex County Hospital, Brighton, United Kingdom

REFERENCES:
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Seupaul RA, Wilbur LG. Evidence-based emergency medicine. Does therapeutic hypothermia benefit survivors of cardiac arrest? Ann Emerg Med. 2011 Sep;58(3):282-3. doi: 10.1016/j.annemergmed.2011.02.002. Epub 2011 Mar 24. No abstract available. PMID 21435740
- See also: Our study location. — http://www.bsms.ac.uk/research/ciru/
- See also: UK health regulatory authority. — http://www.hra.nhs.uk/
- See also: The UK MHRA. — http://www.mhra.gov.uk/Aboutus/index.htm